CLINICAL TRIAL: NCT00722891
Title: Ocular Responses to Acute and Chronic Lens Wear
Brief Title: Ocular Responses to Short and Long-term Lens Wear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: P/289/07/B
Record Dates: First submitted 2008-07-24; First posted 2008-07-28 (Estimated); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Ametropia
Keywords: Eye Diseases
MeSH Terms: conditions — Refractive Errors; Eye Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Purevision Lens with ReNu (Active Comparator): Purevision Lenses with ReNu Multiplus Solution
  Interventions: Device: Purevision Lenses with ReNu Multiplus
- Purevision Lenses with RepleniSH (Active Comparator): Purevision Lenses with Optifree RepleniSH Solution
  Interventions: Device: Purevision Lenses with Optifree RepleniSH

INTERVENTIONS:
Device: Purevision Lenses with ReNu Multiplus — Purevision lenses using ReNu Multiplus lens solution for 28 days
  Other Names: Balafilcon A
  Arms: Purevision Lens with ReNu
Device: Purevision Lenses with Optifree RepleniSH — Purevision lenses using Optifree RepleniSH lens solution for 28 days
  Other Names: Balafilcon A
  Arms: Purevision Lenses with RepleniSH

SUMMARY:
The purpose of this study was to determine whether ocular surface sensitivity to pneumatic, mechanical and chemical stimulation would be affected by the use of the combination of a specific silicone hydrogel lens material with two lens care products over a four week period.

ELIGIBILITY:
Inclusion Criteria:

* Is at least 17 years old and has full legal capacity to volunteer;
* Is correctable to a visual acuity of 6/7.5 (20/25) or better (both eyes) with their habitual vision correction;
* Is a current soft lens wearer and wears contact lenses six or more days/week;
* Has clear corneas and no active ocular disease.

Exclusion Criteria:

* Has any clinically significant blepharitis or dry eye;
* Has undergone corneal refractive surgery;
* Is aphakic;
* Has any active ocular disease;
* Has any systemic disease affecting ocular health;
* Is using any systemic or topical medications that may affect ocular health;

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-07; Primary Completion 2009-06 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Quantify the ocular response to acute and chronic lens wear using slit lamp examination, tear assay and corneal sensitivity. | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Trefford Simpson, DipOptom,MSc,PhD, Principal Investigator — University of Waterloo
Locations (1):
- University of Waterloo, Waterloo, Ontario, Canada